CLINICAL TRIAL: NCT02323074
Title: Brain Training System Using Electroencephalography (EEG) for Neurorehabilitation of Hand Function After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUHK 525513
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- fBCI-robot (Experimental): focalized BCI-robot hand training
  Interventions: Procedure: Brain Computer Interface
- gBCI-robot (Experimental): generalized BCI-robot hand training
  Interventions: Procedure: Brain Computer Interface
- sham-BCI (Sham Comparator): Sham BCI
  Interventions: Procedure: Brain Computer Interface

INTERVENTIONS:
Procedure: Brain Computer Interface

SUMMARY:
In this project we will design a control algorithm to identify the focalized motor-related clusters for hand function on each stroke patient. A real-time feedback will control the robotic hand when motor imagery is successfully identified. Finally, the focalized BCI-robot training will be compared in a randomized controlled trial to evaluate the training effectiveness and changes in the EEG patterns.

ELIGIBILITY:
Inclusion Criteria:

(1) sufficient cognition to follow simple instructions, as well as understand the content and purpose of the experiment (Mini-Mental State Examination (MMSE) score>25) ; (2) subcortical location of the ischemic lesion within the territory of the middle cerebral artery; (3) have moderate to severe motor disability at the paretic upper limb (assessed by Fugl-Meyer Assessment (FMA), Modified Ashworth Score of fingers (MAS), and Action Research Arm Test (ARAT))

Exclusion Criteria:

(1) severe hand spasticity, open hand wound or hand deformity; (2) visual field deficits; (3) aphasia, neglect, and apraxia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
FMA-UE | 3-month followup

SECONDARY OUTCOMES:
ARAT | 3-month followup
MAS | 3-month followup

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Biomedical Engineering, Dept Electronic Engineering, Hong Kong, Hong Kong